CLINICAL TRIAL: NCT06574230
Title: Effect of Regular Dart Training on Visual Perception and Attention Level in Pre-school Children
Brief Title: Dart Training Effect on Visual Perception and Attention Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate Professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/01-09
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Preschool Children; Healthy
Keywords: exercise; dart training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dart training (Experimental): The exercise group participated in dart training for 12 weeks, with sessions held three times per week, each lasting 90 minutes. During the first week of the program, participants received both theoretical and practical instruction on game rules, breathing techniques, and throwing techniques. The training focused on breathing control, throwing techniques, scoring strategies, and involved practicing a set number of exercises.
  Interventions: Other: TRAINING PROGRAM
- control group (No Intervention): the control group did not engage in any dart-related activities during this period and were instructed to continue with their regular daily activities at school.

INTERVENTIONS:
Other: TRAINING PROGRAM — Each training session included a structured set of exercises aimed at enhancing these skills. For example, participants practiced precision drills to target specific areas of the dartboard, endurance drills to build stamina for longer games, and competitive exercises to simulate real-game conditions. This combination of theoretical knowledge, practical skill development, and strategic gameplay was designed to comprehensively improve the participants' dart-throwing abilities over the course of the program. A 12-week dart training program, with sessions conducted three times per week, each lasting 90 minutes. In the first week, participants received comprehensive theoretical and practical instruction covering the rules of the game, proper breathing techniques, and throwing mechanics. This initial phase was designed to ensure a solid understanding of the fundamentals before progressing to more advanced training.
  Arms: dart training

SUMMARY:
Engagement in structured physical and sports activities is widely recognized as an effective method for enhancing visual perception and attention levels. Studies have demonstrated that dart training, in particular, has a beneficial effect on visual perception and attention. Research consistently underscores the significance of visual perception and attention in the accuracy of dart throwing. As dart training enhances these cognitive functions, the integration of visual perception and attention-focused instructions has been shown to improve throwing accuracy. However, the existing literature on this topic, especially regarding pre-adolescent populations, remains limited. Furthermore, evaluating the impact of a structured dart exercise program on both attention and visual perception simultaneously is considered a crucial factor that underscores the significance of this research. This study aimed to determine the effects of dart exercises on the visual perception and attention parameters of pre-adolescent students.

The study included 45 preschool children, with 23 in the experimental group (12 girls and 11 boys) and 22 in the control group (11 girls and 11 boys). Baseline testing of attention and visual perception was conducted prior to the start of the structured dart exercise program, which lasted for 12 weeks. The exercises were performed three days a week, with each session lasting 90 minutes. After 12 weeks, visual perception and d2 attention tests were administered to both the exercise and control groups.

DETAILED DESCRIPTION:
The relationship between dart training and cognitive function has been well-documented. Studies have consistently demonstrated that visual perception and attention are critical for dart-throwing accuracy, and that structured dart training can improve these skills. Moreover, the inclusion of exercises specifically designed to target visual perception and attention has been shown to further enhance throwing accuracy, highlighting the importance of integrating cognitive training with physical practice.

Despite the promising findings, there is a noticeable gap in the literature, particularly concerning the pre-adolescent population. Few studies have explored the effects of dart training on visual perception and attention in this age group. Additionally, there is a lack of research that simultaneously evaluates the impact of a structured dart exercise program on both attention and visual perception, which is crucial for understanding the comprehensive benefits of such interventions.

To address this gap, the present study aimed to assess the effects of dart exercises on the visual perception and attention parameters of pre-adolescent students. The study included 45 preschool children, divided into an experimental group (23 children: 12 girls and 11 boys) and a control group (22 children: 11 girls and 11 boys). Baseline assessments of attention and visual perception were conducted prior to the intervention. The structured dart exercise program, which spanned 12 weeks, consisted of sessions held three days a week, each lasting 90 minutes. Following the completion of the program, visual perception and d2 attention tests were administered to both the experimental and control groups to evaluate the impact of the dart exercises.

ELIGIBILITY:
Inclusion Criteria:

* secondary school students
* being a 5th grade students
* never been playing darts before

Exclusion Criteria:

* having any cardiovascular, neurological, orthopedic, or psychiatric disease
* students who are not taking any regular medication.

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-02-12 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Visual Perception Test | From enrollment to the end of treatment at 12 weeks
  The test includes 13 multiple-choice questions. Each question had four options. The test duration was approximately 30 min, and the tests were performed individually. The evaluation of the test is made out of a total of 100 points, with 7.69 points given for each correctly answered question. Therefore, the lowest score that could be obtained from the test was 0, and the highest score was 100. As the score obtained from the test increased, students' visual perception skills increased.
Attention Test | From enrollment to the end of treatment at 12 weeks
  The attention Test measures selective attention and mental concentration over time. The test can be applied individually or in groups to individuals between the ages of 9-60. The one-page test form contained 14 rows, 47 in each row, for a total of 658 figures. The letters d and p are used in the test. Some letters have one, two, three, or four dots above or below them. In the test, letters can be found in 16 different ways, depending on where they take the dots and their numbers. The main task of the person taking the test was to find the letter d, which had a total of two dots. These can be observed in the tests in three different ways. The test taker had 20 seconds to perform the task specified in each row. The test completion time was approximately eight minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Çalık Veli KOÇAK, PhD, Principal Investigator — Aksaray University

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data might not be shared due to concerns about privacy and confidentiality, especially when dealing with sensitive information that could potentially identify participants.